CLINICAL TRIAL: NCT01771744
Title: Revisional Versus Primary Roux-en-Y Gastric Bypass: a Case Matched Analysis
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Tarik Delko, Dr, University Hospital, Basel, Switzerland
Other Study IDs: Revisional Limmi 1
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Effect of Revisional Surgery for Failed Gastric Banding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Morbidly obese patients: 48 morbidly obese patients with revisional gastric bypass
- 48 morbidly obese patients: with primary gastric bypass

SUMMARY:
This study compared revisional malabsorptive laparoscopic very very long limb gastric bypass (VVLL RYGB) with primary VVLL RYGB and tested the hypothesis that one staged revisional laparoscopic VVLL RYGB is a safe and effective procedure after failed restrictive gastric banding.

ELIGIBILITY:
Inclusion Criteria:

* Primary Gastric Bypass according to SMOB (Swiss group for the study of morbid obesity) Guidelines
* Revisional Gastric Bypass after failed Gastric Banding

Exclusion Criteria:

* According to SMOB Criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: morbidly obese patients
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2000-01; Primary Completion 2010-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
weight loss | 2 years

SECONDARY OUTCOMES:
Complication rate | early (30 days) and late (> 30 days)